CLINICAL TRIAL: NCT01472549
Title: Antiseptic Skin Preparation for Preventing Surgical Site Infection at Cesarean Delivery: a Randomized Comparative Effectiveness Trial
Brief Title: The Skin Prep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB ID #: 201105161
Record Dates: First submitted 2011-09-20; First posted 2011-11-16 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Surgical Site Infections
Keywords: Preoperative; Antiseptics; Comparative; Cost; Effectiveness
MeSH Terms: conditions — Surgical Wound Infection | interventions — Iodine; Ethanol; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodine-alcohol (Active Comparator): 8.3% povidone-iodine with 72.5% alcohol (Prevail-FX, Cardinal Health)
  Interventions: Drug: Iodine-alcohol
- Chlorhexidine-alcohol (Experimental): 2% chlorhexidine gluconate with 70% alcohol (ChloraPrep, Cardinal Health)
  Interventions: Drug: Chlorhexidine-alcohol

INTERVENTIONS:
Drug: Iodine-alcohol — Skin preparation with 8.3% povidone-iodine with 72.5% alcohol (Prevail-FX, Cardinal Health) preoperative skin preparation.
  Other Names: Prevail-FX, Cardinal Health
  Arms: Iodine-alcohol
Drug: Chlorhexidine-alcohol — Skin preparation with 2% chlorhexidine gluconate with 70% alcohol (ChloraPrep, Cardinal Health) preoperative skin preparation
  Other Names: ChloraPrep, Cardinal Health
  Arms: Chlorhexidine-alcohol

SUMMARY:
The investigators propose a randomized controlled clinical trial to determine the comparative effectiveness of chlorhexidine-alcohol and iodine-alcohol preoperative skin preparation for preventing surgical site infections at cesarean section. While estimates vary, surgical site infections complicate up to 5 - 10% of all cesarean sections and result in significant human suffering and excess health care costs. Interventions such as preoperative antibiotic prophylaxis reduce surgical site infections by 60%, but the rate of infection remains high. There is therefore a great need to identify and test other potential interventions to further reduce these infections.

The skin is a major source of pathogens that cause surgical site infection. Therefore, optimizing preoperative skin antisepsis has the potential to decrease postoperative surgical site infections. There is paucity of evidence to guide the choice of antiseptic for skin preparation at cesarean section. To date, only two underpowered trials have been published comparing two methods of preoperative skin preparation at cesarean section. A recent randomized trial in adults undergoing clean-contaminated mostly general surgical procedures demonstrated a 41% reduction in surgical site infection with the use of chlorhexidine-alcohol when compared to the more commonly used povidone-iodine. While it is plausible that findings from trials in other clean-contaminated surgical procedures may apply to cesarean sections, physiological changes in pregnancy, the peculiar dual microbial source for cesarean-related infections and the hormone-mediated immune-modulation in pregnancy make the validity of such extrapolation uncertain.

The study has the following specific aims:

Primary Aim: To test the hypothesis that preoperative chlorhexidine-alcohol skin preparation at cesarean section significantly reduces surgical site infections compared to iodine-alcohol.

Secondary Aim 1: To test the hypothesis that preoperative chlorhexidine-alcohol skin preparation at cesarean section significantly reduces bacterial contamination at the surgical site compared to iodine-alcohol.

Secondary Aim 2: To determine clinical outcomes and medical costs associated with cesarean-related infections and quantify potential cost savings attributable to use of chlorhexidine-alcohol for preoperative skin preparation at cesarean section.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

This will be a randomized controlled clinical trial aimed at determining the comparative effectiveness of chlorhexidine-alcohol and iodine-alcohol preoperative skin preparation for preventing surgical site infection at cesarean section.

The investigators will use broad inclusion criteria and analyze all the main outcomes by the intent-to-treat principle. This approach will allow a more conservative estimate of differences between groups and allow a better estimate of effectiveness and public health implications of practice change rather than a pure estimate of efficacy alone.

Randomization and Treatment: Enrolled patients will be randomly assigned in a 1:1 ratio using computer-generated randomization sequence to the two skin preparation methods.

Blinding: Blinding both patients and physicians to the antiseptic used for skin preparation (double-blinding) would be ideal. However, it is not feasible in this trial. First, most patients can determine whether they were assigned to chlorhexidine or iodine, as the two antiseptics are of different colors and leave a stain on the skin (pink or brown, respectively). Second, physicians are often in the operating room when the skin is being prepared for cesarean section and will know which antiseptic is used. We will minimize systematic bias by using the same standard procedures of skin preparation, skin culture and assessment of outcomes. All diagnoses of surgical site infection will be verified by chart review using the Centers for Disease Control and Prevention (CDC) National Nosocomial Infections Surveillance System criteria. The principal investigator will verify the diagnoses without knowledge of the group to which the patients were assigned.

PRIMARY AIM:

Outcome measures-Primary outcome-Proportion of subjects with surgical site infection (superficial incisional [skin, subcutaneous layer] or deep incisional [fascia, muscle]) within 30 days of cesarean delivery. Surgical site infection will be based on diagnosis by the treating physician and verified by chart review in accordance with the CDC Nosocomial Infections Surveillance System definitions.

Secondary outcomes-Length of hospital stay, number of office visits and re-admissions for infection-related complications, endometritis, positive culture from wound culture, skin irritation and allergic reactions.

Methods-Subjects will undergo cesarean delivery based on the technique selected by the surgeon. The circulating nurse will record information on key variables known to be related to surgical site infection: antibiotic administration (type and timing), type of cesarean section (scheduled or emergent), status of membranes (ruptured or unruptured), duration of surgery, depth of subcutaneous layer (closed or not closed) and skin closure method (subcuticular suture or staples) on data collection forms.

Demographic (age, race, socioeconomic status), obstetric (parity, gestational age, indication for cesarean section, cervical dilation at time of cesarean section, presence of chorioamnionitis, surgical complications) and neonatal (birth weight, Apgar score, cord pH) data will be abstracted from the patients chart.

Subjects will be contacted once, up to 30 days from delivery, to assess symptoms of cesarean-related infections. Patients who report symptoms will be directed to follow up in the emergency department or with their physician to be evaluated for surgical site infection. Wound swabs will be taken for aerobic and anaerobic cultures in all subjects who present at Barnes-Jewish Hospital with wound infection. Medical records will be obtained from treating physicians to determine the diagnosis at each postoperative office visit or readmission within 30 days of cesarean section.

Statistical Analysis: Data analyses will be based on the intent-to-treat principle. The primary outcome (proportion of subjects with surgical site infection) and the other categorical variables will be compared across groups using the chi-squared test. Fisher's exact test will be used for variables in which expected numbers in any of the cells in 2 x 2 tables is <5. We will calculate 95% confidence intervals around the differences in proportions and the relative risk of surgical site infection.

Distribution of continuous variables will be evaluated by visual inspection of histograms and the Kolmogorov-smirnov test. Normally distributed variables will be compared using the unpaired t-tests. If variables are not normally distributed, log transformation will be used in an attempt to achieve normal distribution. If the data is still skewed after log transformation the Mann-Whitney U test will be used to compare groups.

It is anticipated that baseline characteristics will be similar in the two groups. In the event that the groups are unbalanced with regards to variables significantly associated with the primary outcome, supplemental analyses will be performed using stratification on the individual variables and multivariable logistic regression adjusting for multiple covariates.

Planned subgroup analysis will be performed for: i. scheduled and elective cesarean sections, iii. obese and normal weight women, iii. Subcuticular and staple closure, and iv. women with and without chronic medical conditions (diabetes, chronic hypertension, renal disease). Interaction tests will be used to determine if the effectiveness of the skin preparation methods differ across these subgroups. Tests with p <0.05 will be considered statistically significant. Analyses will be performed using Stata version 10.0 (Stata Corp., College Station, TX).

Sample Size Estimation: The sample size estimation for the primary aim is based on an assumed baseline surgical site infection rate of 8% and an anticipated clinically significant 50% reduction in surgical site infection. To have 80% power to detect 50% difference in a two-tailed chi-squared test with α of 0.05, a total of 1084 subjects will need to be randomized. To accommodate a 10% drop out rate, 1, 192 subjects will be enrolled (596 chlorhexidine, 596 iodine).

SECONDARY AIM #1:

To test the hypothesis that preoperative chlorhexidine-alcohol skin preparation at cesarean section significantly reduces bacterial contamination at the surgical site compared to povidone-iodine Primary outcome-Proportion of subjects with surgical site skin contamination after antiseptic preparation. Contamination will be defined as ≥5000 total colony-forming units per milliliter on aerobic or anaerobic culture.

Secondary outcomes-Types of bacteria cultured before and after skin preparation, concordance of bacteria at surgical site following preoperative skin preparation with bacteria in postoperative surgical site infections.

Methods-Two skin swabs will be taken transversely across the suprapubic area, 2 finger breadths above the symphysis pubis immediately before, and 5 minutes after skin preparation. These swabs will be cultured under aerobic and anaerobic conditions. To ensure that the groups at high risk for surgical site infections are well represented, we will ensure that obese women, diabetics and women undergoing emergent cesarean deliveries are adequately sample and randomized.

Statistical Analysis-Data analyses will be based on the intent-to-treat principle. The primary outcome (proportion of subjects with surgical site skin contamination after skin preparation) and the other categorical variables will be compared across groups using the chi-squared test. Fisher's exact test will be used for variables in which expected numbers in any of the cells in 2 x 2 tables is <5. Tests with p <0.05 will be considered significant. We will also conduct stratified analysis based on the different risk groups. Finally, we will calculate 95% confidence intervals around the difference in proportions and relative risk of skin contamination after antiseptic skin preparation. Analyses will be performed using Stata version 11.0 (Stata Corp., College Station, TX).

Sample Size Estimation-The sample size estimation for secondary aim #1 is based on the primary outcome of skin contamination following skin preparation. A meta-analysis of data from non-obstetric surgical procedures suggest a contamination rate of 39% after preoperative skin preparation with iodine and a rate of 18% after the use of chlorhexidine [17]. On the basis of an assumed contamination rate of 39% in the iodine group and 50% difference in skin contamination as clinically significant, a total of 168 subjects will be needed (84 chlorhexidine, 84 iodine) to have 80% power in a two-tailed chi-squared test and α of 0.05.

SECONDARY AIM #2 The outcome for secondary aim#2 is attributable cost saving (if any), defined as the difference in total costs between women with preoperative iodine and chlorhexidine skin preparation.

Methods/Data Analysis-A cost-benefit decision analysis model will be developed depicting the decision of whether to use chlorhexidine or iodine for a patient undergoing cesarean section. The cost of implementing each strategy will include the purchase costs of the antiseptic agents. For each antisepsis strategy, the patient would then have a probability of subsequently developing surgical site infection based on results of the randomized trial under the primary aim. We will calculate cost incurred by patients who did and did not develop an infection.

Costs will be obtained from the Barnes-Jewish Hospital cost accounting database for the surgical admission and any readmission to the hospital and office visits within 30 days after cesarean section. Cost savings, if any, will be the difference between the costs in the two groups. The cost-benefit analysis will be performed using TreeAge Pro 2009 (TreeAge Software).

Sample Size Estimation-No formal sample size estimation is made for secondary aim #2. The cost-benefit analysis will be based on outcomes among the subjects enrolled under secondary aim #2.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean delivery at Barnes-Jewish Hospital.

Exclusion Criteria:

* Inability to obtain consent; allergy to chlorhexidine, alcohol, iodine, shellfish; and evidence of infection adjacent to operative site.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Methodius G Tuuli, MD, MPH, Principal Investigator — Washington University School of Medicine; George Macones, MD, MSCE, Study Chair — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tuuli MG, Liu J, Stout MJ, Martin S, Cahill AG, Odibo AO, Colditz GA, Macones GA. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. N Engl J Med. 2016 Feb 18;374(7):647-55. doi: 10.1056/NEJMoa1511048. Epub 2016 Feb 4. PMID 26844840
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this single-center, randomized, controlled trial, a total of 1147 patients were enrolled from September 2011 through June 2015.
Period: Overall Study
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Started | 572 | 575
Completed | 572 | 575
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol | Total
Number analyzed (Participants) | 572 | 575 | 1147
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.8) | 28.4 (5.8) | 28.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 572 | 575 | 1147
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 572 | 575 | 1147
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 35.1 (8.9) | 34.1 (8.1) | 34.6 (8.5)
Scheduled cesarean [Count of Participants; unit: Participants] | 334 | 335 | 669

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infection
Description: Superficial or deep surgical-site infection within 30 days after cesarean delivery, on the basis of the National Healthcare Safety Network definitions of the Centers for Disease Control and Prevention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
Participants | 23 | 42
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.55, 95% CI 2-sided [0.34 to 0.90]

2. Secondary Outcome: Length of Hospital Stay
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
days | 4 [3 to 4] | 4 [3 to 4]
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants With Re-admissions or Office Visits for Wound-related Problems
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
Participants | 19 | 25
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.43 to 1.37]

4. Secondary Outcome: Number of Participants With Endometritis
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
Participants | 8 | 11
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.49, Chi-squared; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.30 to 1.80]

5. Secondary Outcome: Number of Participants With Skin Irritation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
Participants | 0 | 3
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.08, Fisher Exact

6. Secondary Outcome: Number of Participants With Allergic Reaction
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 572 | 575
Participants | 2 | 1
Statistical Analysis 1: Comparison: Chlorhexidine-alcohol vs Iodine-alcohol; Test type: Superiority; p = 0.56, Fisher Exact; Risk Ratio (RR) = 2.02, 95% CI 2-sided [0.18 to 22.11]

7. Secondary Outcome: Number of Participants With Skin Contamination After Skin Prep
Time Frame: 1 day
Population: The skin samples collected could not be processed for financial reasons.
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 00000 | 00000

8. Secondary Outcome: Cost Savings
Time Frame: 30 days
Population: Cost data was not collected because it as not logistically feasible.
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
Number analyzed (Participants) | 00000 | 00000

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Chlorhexidine-alcohol | Iodine-alcohol
All-Cause Mortality (participants affected / at risk) | 0/572 | 0/575
Serious Adverse Events (participants affected / at risk) | 0/572 | 0/575
Other Adverse Events (participants affected / at risk) | 15/572 | 15/575
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine-alcohol (N=572) | Iodine-alcohol (N=575)
Adverse skin reactions (Skin and subcutaneous tissue disorders) | 15 (15) | 15 (15) — Adverse skin reactions including erythema, skin irritation and allergic skin reactions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes